CLINICAL TRIAL: NCT01573533
Title: A Pilot Study to Assess the Efficacy of Rituximab Therapy in Patients With Treatment Resistant Idiopathic Focal Segmental Glomerulosclerosis (FSGS): Integrating an Assessment of the Relevance of suPAR and Activation of Podocyte β3 Integrin
Brief Title: A Pilot Study to Assess the Efficacy of Rituximab Therapy in Treatment Resistant FSGS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University Health Network, Toronto (Other); National Institutes of Health (NIH) (NIH); Genentech, Inc. (Industry); Rush University Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Fernando Fervenza, PI, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-005640; U54DK083912 (NIH)
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Primary Focal Segmental Glomerulosclerosis
Keywords: Treatment Resistant Idiopathic FSGS; Glomerulosclerosis; Proteinuria; Rituximab
MeSH Terms: conditions — Proteinuria | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab (Experimental)
  Interventions: Biological: Rituximab

INTERVENTIONS:
Biological: Rituximab — Rituximab will be infused intravenously on Day 1 and Day 15 at a dose of 375 mg/m2 up to a maximum of 1000mg per dose in children and at a dose of 1000 mg on Day 1 and Day 15 in adults.
  Other Names: Rituxan®

SUMMARY:
The purpose of this study is to determine whether Rituximab therapy is safe and effective in treating patients with the kidney condition, focal segmental glomerulosclerosis (FSGS), that is no longer responsive to traditional therapies.

DETAILED DESCRIPTION:
This is a pilot trial to assess the safety, feasibility and efficacy of Rituximab therapy in 20 adult and pediatric patients with either steroid and/or calcineurin inhibitor resistant FSGS or with a significant intolerance or contraindication to the use of these agents. In addition to clinical criteria, elevated levels of suPAR will define inclusion. Changes in the baseline levels of the potential biomarkers (suPAR, as well as activation of beta-3 integrin) in response to treatment will be compared to clinical measures of efficacy.

Participants will have a screening/baseline visit to confirm eligibility within 6 weeks prior to the first of two Rituximab infusions (at Day 1 and Day 15). Participants will then attend follow up visits at 1, 3, 6 and 12 months after Rituximab treatment to assess adverse events and collect safety blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* FSGS involving native kidneys with a diagnostic biopsy performed within the last 3 years
* Patients >6 years of age and < 80 years of age
* suPAR > 3500 pg ml-1
* Treatment with an ACEI and/or ARB as tolerated for at least 3 months prior to enrollment to with a target a systolic blood pressure ≤ 140 mmHg and a diastolic pressure ≤ 90 mmHg in adults and blood pressure readings less than the 95th percentile for age, gender and height in children in at least 75% of readings
* Proteinuria ≥ 3.0 grams as measured by 24-hour urine collection in adults and urine protein:creatinine ratio ≥ 1.0 in the first morning urine in children, despite ACE inhibitor / ARB treatment as tolerated and a minimum of 8 weeks of prednisone therapy at ≥ 1 mg/kg/day, a trial of calcineurin inhibitor for=> 3 months or a contraindication/intolerance to such therapy (diabetes, osteoporosis/osteonecrosis, age >60, BMI ≥35)
* Negative serum pregnancy test (for women of child bearing age)
* Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of the trial
* Able and willing to give written informed consent and comply with study requirements

Exclusion Criteria:

* Estimated GFR < 40 ml/min per1.73m2. The rationale is that patients with advanced renal failure may progress rapidly towards ESRD.
* Collapsing variant of FSGS, as it is rare and has been associated with an aggressive course
* Concurrent use of immunosuppressive therapy with the exceptions of prednisone 10 mg/day. Patients who are taking other immunosuppressive therapy, must be off immunosuppressive medications for equal to or > 3 months prior to enrollment into the study with the exception of patients demonstrating significant worsening of proteinuria (of >30% above baseline) during the washout period. These resistant patients can be treated after 1 month of washout due to the high likelihood of progression and/or lack of delayed (previous) immunosuppression effect.
* Patients with medical conditions that may cause FSGS (e.g. HIV, lymphoma, heroin use) or have a secondary form of FSGS due to hyperfiltration injury (massive obesity, vesicoureteral reflux, or renal mass reduction)
* Type 1 or type 2 diabetes mellitus as diabetic glomerulosclerosis may be contributing to proteinuria in these patients
* History of serious recurrent or chronic infection
* Presence or suspicion of active infection including TB, HIV, Hepatitis B and HCV with positive tests for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis B virus (HBV), Hepatitis C serology, HIV serology or a positive TB skin test, which require further investigation to rule out active disease (ie. chest x-ray)
* Known active infection requiring hospitalization or treatment with intravenous antibiotics within 4 weeks or oral antibiotics within 2 weeks of the study initiation
* Low immunoglobulins (level to be based on age)
* Absolute neutrophil count < 1.5 x103/mL
* Patients in receipt of a live vaccine within 4 weeks of the study initiation
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Previous Treatment with a B-cell depleting antibody
* History of severe allergic reactions to humanized or murine monoclonal antibodies
* Treatment with any investigational agent within 4 weeks of the study initiation
* History of major psychiatric disorder, drug or alcohol abuse within the previous 6 months
* Any other disease, metabolic dysfunction, physical examination finding or clinical laboratory that provides a reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hladunewich, MD, MSc, BSc, Principal Investigator — University Health Network, Sunnybrook Health Sciences Centre; Fernando C Fervenza, MD, PhD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic College of Medicine, Rochester, Minnesota
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1
  Canada | 8

OUTCOME MEASURES:

1. Primary Outcome: Changes in Proteinuria (With Stable Renal Function)
Description: The amount of protein in excreted urine measured by grams per day (g/day). Remission status defined by the following criteria at 12 months:
  * Complete Remission - Proteinuria < 0.5 g/day
  * Partial Remission - Improvement in proteinuria by > 50% and to a level between 0.5-3.5g/day
  * Incomplete Remission - Improvement in proteinuria equal to or >50%, but residual proteinuria still >3.5g/day
Time Frame: Baseline, 12 months
Measure: Mean (Standard Deviation); unit: g/day
Arm/Group | Rituximab
Number analyzed (Participants) | 9
g/day
  Baseline | 7.6 (4.67)
  12 months | 7.27 (7.30)
Statistical Analysis 1: Comparison: Rituximab; Baseline vs 12 months; Test type: Superiority; p = 0.49, ANOVA

2. Secondary Outcome: Change in suPAR Levels
Description: SuPAR concentrations will be determined by quantitative ELISA immunoassay reported in picograms per milliliters (pg/ml)
Time Frame: Baseline, 1, 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Rituximab
Number analyzed (Participants) | 9
pg/ml
  Baseline | 4120 (1169)
  1 month | 3730 (1229)
  3 month | 4231 (1871)
  6 month | 4491 (2217)
  12 month | 3788 (1836)
Statistical Analysis 1: Comparison: Rituximab; Baseline vs 12 months; Test type: Superiority; p = 0.41, ANOVA

3. Secondary Outcome: Change in Activation of Podocyte β3 Integrin
Description: To quantitatively examine the effect of FSGS patient sera on podocyte β3 integrin activity, a human podocyte cell line is cultured at 37 degrees Celsius for 14 days for complete differentiation. The cells are then incubated in 5-10% of FSGS patient serum for 24 hours with recombinant suPAR protein as a positive control. Cells are fixed with 4% paraformaldehyde (PFA) and proceeded for immunofluorescence staining for AP5 and paxillin. After immunostaining, confocal images are taken to quantify the AP5 and paxillin intensity for each sample treatment. Paxillin signal is used to correct AP5 signal. The relative AP5 signal (AP5/paxillin ratio) from each patient serum is then normalized against that of normal blood donor included in each assay for final report.
Time Frame: Baseline, 1, 3, 6, 12 months
Measure: Mean (Standard Deviation); unit: AP5/paxillin ratio
Arm/Group | Rituximab
Number analyzed (Participants) | 9
AP5/paxillin ratio
  Baseline | 1.56 (0.59)
  1 month | 1.17 (0.17)
  3 month | 1.13 (0.34)
  6 month | 1.15 (0.30)
  12 month | 1.24 (0.27)
Statistical Analysis 1: Comparison: Rituximab; Baseline vs 12 months; Test type: Superiority; p = 0.06, ANOVA

4. Secondary Outcome: Number of Subjects With Complete or Partial Remission Following Treatment
Description: Total number of subjects with complete or partial remission following treatment using the following criteria:
  * Complete Remission - Proteinuria < 0.5 g/day
  * Partial Remission - Improvement in proteinuria by > 50% and to a level between 0.5-3.5g/day
  * Incomplete Remission - Improvement in proteinuria equal to or >50%, but residual proteinuria still >3.5g/day
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: The study period during which all AEs and SAEs must be reported begins after informed consent is obtained and ends 30 days after study discontinuation/termination for each participant.
Arm/Group | Rituximab
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=9)
Lung Infection (Infections and infestations) | 1 (1)
Acute Kidney Infection (Renal and urinary disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=9)
Relapse of Nephrotic Syndrome (Renal and urinary disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Sore Throat (General disorders) | 1 (1)
Cramps (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Weakness (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Rash (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Nail Infection (Infections and infestations) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT01573533/Prot_SAP_000.pdf